CLINICAL TRIAL: NCT04731311
Title: Telerehabilitation Combining Virtual Reality Adaptable Games and Drug Therapy for Early Alzheimer's Disease - Usability
Brief Title: Telerehabilitation Alzheimer's Disease Usability (TADU)
Acronym: TADU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bright Cloud International Corp (Industry)
Collaborators: National Institute on Aging (NIA) (NIH); Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Telerehab AD Usability; R43AG065035 (NIH)
Record Dates: First submitted 2021-01-23; First posted 2021-01-29 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Alzheimer Disease; Healthy Aging
Keywords: Alzheimer's Disease; Virtual Reality; BrightGo; Head Mounted Display; Aricept; Exelon
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: All participants will perform same protocol consisting of 4 evaluation sessions of the BrightGo device
Masking Description: No Masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Usability Evaluation of the BrightGo system (Other): Participants with rate the device in each of 4 usability evaluation sessions.
  Interventions: Device: Usability evaluation of BrightGo computerized device for cognitive therapy of individuals with early Alzheimer's Disease

INTERVENTIONS:
Device: Usability evaluation of BrightGo computerized device for cognitive therapy of individuals with early Alzheimer's Disease — 4 participants with undergo 4 usability evaluations each, inter-spaced by days when researchers will address design changes. 2 participants will be elderly healthy and 2 will have the early Alzheimer's disease. Each session will last up to 1 hour, during which participants will interact with tasks in the form of games. Games will be gradated in level of difficulty, increasing from session to session. They will be played with one game controller or with two controllers while participants wear an all-in-one head mounted display. The degree of cognitive engagement during tasks will be measured with custom biosensors and used in adjusting level of difficulty. Each participant will fill subjective evaluation form and a USE form assessing ease of use, usefulness, and perceived technology issues. Scores will be analyzed and data published, in conjunction with game performance data.

SUMMARY:
Usability evaluation of BrightGo cognitive telerehabilitation system. An experimental system was developed to enhance standard of care (medication effect) for Early Alzheimer's Disease populations. This computerized system will be undergo a usability evaluation by healthy and by elderly participants who are in the early phase of Alzheimer's Disease. Sessions will and with participants filling subjective evaluation questionnaires as well as the USE standardized form. Results will be used to address any uncovered issues before a follow on Pilot RCT Feasibility study. Participants will receive $25 after each evaluation session.

DETAILED DESCRIPTION:
Study will start with 2 elderly healthy volunteers (one male and one female) with preference to those with no computer game experience. The healthy volunteers will each perform usability sessions (2 times per week) in the first 2 weeks. They will be instructed to move the arms, grasp and extend fingers, so to mimic the assumed functionality during subsequent feasibility component.

The usability subjects will test the game controller movement, the caregiver tablet interface, and test all therapeutic games. Each of the games will be tested at all levels of difficulty, so to detect any previously unknown bugs. They will further test system wireless communication and real-time graphics response to controller input (minimal lag and lack of freezing, smooth avatar control). Finally, they will test the set motor and cognitive baseline procedures, meant to adapt games to participant. Specifically, this research team has developed a relaxing scene to be shown to participants while their biosensors are measured. This will help interpret any changes occurring subsequently, during therapeutic game interactions so to get an indication of engagement, or lack of, with the game tasks.

At the end of each session, volunteers will fill in the USE standardized usability questionnaire [Lund 2001]. This questionnaire will rate the usefulness, ease of use, ease of learning, and satisfaction with the BrightGo system. The USE form will solicit comments on games instructions, ergonomic issues with the new hand controllers, and degree of assistance needed. Sessions will be inter-spaced with days when the programmer, engineer and our Research Therapist will address issues uncovered in the previous session(s).

The usability evaluation process will be repeated in the subsequent 2 weeks with two participants in the early phase of Alzheimer's disease. Their performance will be compared with that of the elderly healthy volunteers, so to better gauge the usability of the BrightGo system for the targeted population. The Usability study will inform necessary BrightGo system improvements prior to feasibility study. Participants with early phase of Alzheimer's disease will not test the caregiver tablet. Usability participants will be paid $25/session.

ELIGIBILITY:
Inclusion Criteria for healthy volunteers:

* Good or corrected hearing;
* Good or corrected vision;
* No motor or cognitive impairments;
* English speaker;
* Willing to travel to usability site (NJ Bioscience Center)

Inclusion Criteria for individuals with early Alzheimer's Disease:

* Age 65 to 85;
* Diagnosis of early Alzheimer's (Montreal Cognitive Assessment [MoCA] score of 19-25) [Nasreddine et al 2005].
* English speakers;
* Ability to actively move UE and to flex/extend fingers;
* Stable on Aricept 10 mg daily intake, or Exelon 9.5 mg patch medication
* Able to consent;
* Good or corrected hearing;
* Good or corrected vision;
* Good upper extremity motor function, close to full range of movement of arms and fingers;
* Willing to travel to usability site (NJ Bioscience Center)

Exclusion Criteria:

* Those younger than 65;
* Severe visual impairments or legally blind;
* Severe hearing loss or deafness;
* Uncontrolled hypertension (>190/100 mmHg);
* Severe cognitive delay (MoCA <19);
* non-English speakers;
* Those unable to provide consent;
* Unable to move arms and fingers, or with severe arthritis;
* Severe propensity to simulation sickness;

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
USE questionnaire to assess the usability of a computerized system | At each of 4 evaluation sessions over 1 month from enrollment
  A standardized questionnaire to assess the usefulness, satisfaction and ease of use of the BrightGo system [Lund, 2001] when evaluated by study participants. The form consists of 30 questions, each rated on a 7-point Likert scale (1 worst 7 best). The score range for this form is 30 (min) to 210 (max).
  Participants will also be able to comment in free form on aspects they liked most and least about the device.

SECONDARY OUTCOMES:
Subjective rating questionnaire of the device and therapy | At each of 4 evaluation sessions over 1 month from enrollment
  Participants rate the usefulness, satisfaction issues, and ease of use of the BrightGo system and therapeutic games. Form consists of questions, each rated on a 5-point Likert scale (1 worst to 7 best).

OTHER OUTCOMES:
Simulation Sickness Questionnaire for participant | at enrollment (20 minutes)
  Form used at screening post-consent to determine a participant's propensity for simulation sickness [Kennedy et al.,1993]. The questionnaire asks participants to score 16 symptoms on a four point scale (0-3). Score range is 0 (best outcome - no likelihood of experiencing simulation sickness with the device) to 48 (worst outcome - certainty participant will experience severe simulation sickness).
Montreal Cognitive Assessment (MoCA) to measure level of cognitive impairment | at enrollment (20 minutes)
  Used at screening post-consent to determine level of cognitive impairment [Nasreddine et al 2005] for participants. The form has a score range from 0 (worst) to 30 (best) - no cognitive impairments. For the participants with early Alzheimer's Disease the form will confirm the participant is in the score range of 19-25.
Pulse | Before and after each of 4 sessions, over one month from enrollment
  Heart rate measured with medical meter
Blood pressure | Before and after each of 4 sessions, over one month from enrollment
  Systolic and Diastolic blood pressure will be measured with medical meter

CONTACTS AND LOCATIONS:
Overall Officials: Grigore C Burdea, PhD, Principal Investigator — Bright Cloud International Corp
Locations (1):
- Bright Cloud Int'l Corp, North Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
We will not disclose data on individual participants

REFERENCES:
- See also: BCI's corporate site showing therapeutic games used with the device — http://www.BrightBrainer.com